CLINICAL TRIAL: NCT07046429
Title: Effect of Supplemental Nightly Melatonin On REM and Cognition in Hepatic Encephalopathy (SNORE-HE) Trial
Brief Title: Affect of Melatonin on Sleep and Cognition in Cirrhosis
Acronym: SNORE-HE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: American Association for the Study of Liver Diseases (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 25-01028397; TRA25-218891 (Other Grant/Funding Number: American Association for the Study of Liver Diseases)
Record Dates: First submitted 2025-06-23; First posted 2025-07-01 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Hepatic Encephalopathy; Covert Hepatic Encephalopathy; Cirrhosis; Sleep Disturbances and Insomnia
Keywords: cirrhosis; hepatic encephalopathy; covert hepatic encephalopathy; portal hypertension; sleep disturbances; insomnia; sleep problems; wearable technology
MeSH Terms: conditions — Hepatic Encephalopathy; Fibrosis; Parasomnias; Sleep Initiation and Maintenance Disorders; Hypertension, Portal | interventions — Melatonin; Thiamine

STUDY DESIGN:
Intervention Model Description: Sleep is highly complex and individualized. Therefore, it is difficult to properly randomize participants in a small pilot study and then compare sleep physiology ex post facto. Therefore, the investigators will utilize a crossover technique to allow participants to serve as their own controls. Half of participants will be randomized to start with melatonin, and the other half with thiamine. There will be a two week lead in, and there will be a one week crossover washout period.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Melatonin then Thiamine (Experimental): This group will take one month of melatonin, followed by a one week washout period, then one month of thiamine. They will have the primary outcomes assessed at each month, and will also undergo continuous sleep monitoring via a wearable tracker during all phases of the arm.
  Interventions: Dietary Supplement: Melatonin tablet 3 mg once daily; Dietary Supplement: Thiamine
- Thiamine then melatonin (Experimental): This group will take one month of melatonin, followed by a one week washout period, then one month of thiamine. They will have the primary outcomes assessed at each month, and will also undergo continuous sleep monitoring via a wearable tracker during all phases of the arm.
  Interventions: Dietary Supplement: Melatonin tablet 3 mg once daily; Dietary Supplement: Thiamine

INTERVENTIONS:
Dietary Supplement: Melatonin tablet 3 mg once daily — Participants will be instructed to take 3 mg regular acting (not orally dissolving) melatonin 30 minutes before their anticipated bedtime, nightly for the 30 days preceding analysis of study endpoints.
Dietary Supplement: Thiamine — Participants will be instructed to take 100 mg regular acting (not orally dissolving) thiamine 30 minutes before their anticipated bedtime, nightly for the 30 days preceding analysis of study endpoints.

SUMMARY:
The goal of this clinical trial is to learn the affect of melatonin on sleep, cognitive function, and quality of life (QoL) in patients with cirrhosis and a complication called hepatic encephalopathy (HE). The main questions this study aims to answer are:

* Does taking melatonin increase REM sleep, an important part of healthy sleep that is reduced in cirrhosis?
* Does taking melatonin improve cognitive function and reported QoL?

This is a pilot study, where participants will:

* take one month of melatonin, followed by one month of thiamine, which is another supplement but is not suspected to impact sleep significantly.
* Undergo cognitive testing and take surveys
* Wear a commercial wearable sleep tracker
* Have a formal sleep study and salivary melatonin collection at the end of taking each supplement at our sleep center Participants will be blinded, and neither they nor the researchers will know which supplement they are taking first and which they are taking second. They will also be randomized, with half starting with melatonin and the other half starting with thiamine.

DETAILED DESCRIPTION:
Study Objectives

This project aims to determine the impact of melatonin supplementation on sleep physiology in patients with cirrhosis and HE.

Hypothesis: Melatonin supplementation will improve sleep physiology, and REM specifically.

Background and Significance

Hepatic encephalopathy (HE) affects approximately 50% of patients with cirrhosis, causing lasting cognitive and quality of-life impairments even with therapy. Most HE cases are covert, significantly increasing risks of hospitalization, mortality, and progression to overt HE (OHE) within three years (>50%). Guidelines recommend screening all patients for covert HE (CHE) using neurocognitive tools such as the Psychomotor Hepatic Encephalopathy Score (PHES). However, low screening and treatment rates persist due to the need for specialized training, equipment, and significant time commitments. Even in patients receiving HE therapy, clinicians are hesitant to escalate treatment absent overt confusion, largely due to the cost and poor tolerability of rifaximin and lactulose. These limitations contribute to frequent hospital readmissions and high short-term mortality in those with prior OHE. Improved recognition and management strategies are critical to advancing HE outcomes.

Sleep changes in HE are frequently described, often as disturbances in the sleep-wake cycle. The pathophysiology is likely multifactorial, including adenosine mediated hyperammonemic effects on arousal and alterations in endogenous melatonin metabolism in cirrhosis with resultant circadian rhythm dysfunction. Prior research confirms that patients with CHE likewise suffer from suboptimal sleep with associated quality of life reduction, and our research and others have noted reduced REM sleep, and increased sleep fragmentation. There may also be a bi-directional relationship between sleep decline and cognitive impairment in progressive OHE. Traditional gold-standard assessment of sleep physiology utilizes polysomnography (PSG), which requires on-site monitoring, application of multiple cumbersome leads, and costs up to $2000 for a night's study, making it impractical for routine assessment of disturbed sleep in cirrhosis. Consumer wearables have drastically increased in popularity for personal sleep assessment. Their ease of use, affordability, and promising performance in validation studies with PSG make them an attractive target for research. Utilization of wearables in cirrhosis may make sleep a more approachable target for monitoring in CHE. Melatonin is an endogenous pineal hormone with a known role in circadian maintenance with reduced hepatic metabolism and higher baseline serum levels in cirrhosis, perhaps contributing to circadian dysfunction. Prior research suggests that supplementing melatonin in patients with REM sleep disorders, poor subjective sleep, and cirrhosis improves subjective or objective sleep and wellbeing, but have never assessed the impact on cognitive function or CHE. Data suggests melatonin can improve REM sleep duration, sleep latency, and sleep disturbances, while being safe and affordable with high tolerability, but objective data is lacking in cirrhosis and large-scale randomized trials have not been done to date.

Overall Design

This study is a pilot randomized double-blinded, crossover study of melatonin. This design allows participants to serve as their own controls, reducing sample size needed, minimizing inter-individual sleep variability and permitting 1:1 randomization, provided proper washout and analysis for period effect, addressed below. Randomization will be performed in Stata, with a single unblinded coordinator. Each participant will have a 2-week run in for baseline home sleep assessment, 4 weeks on 3 mg nightly melatonin or 100 mg thiamine, a 1-week washout, and a 4-week period on the alternate therapy for a total of 11 weeks in the study. The washout period was chosen from previously published washouts of melatonin. Thiamine was chosen to approximate placebo due to its identical taste/appearance, affordability and lack of hepatotoxicity. After a two-week lead in, the investigational pharmacy will give participants an identical 30-day supply of either 3 mg melatonin tablets or 100 mg thiamine tablets who will be instructed to take it nightly 30-60 min before intended bedtime. A MEDLINE search does not identify any published reports of thiamine impacting melatonin secretion, sleep physiology or sleep quality. Both melatonin and thiamine are dietary supplements and do not require an investigational new drug application (IND) for assessment of sleep physiologic effects. After the first sleep study is completed the bottle will be collected and the alternative therapy will be given, with instructions to start after a one-week washout. Sleep will be tracked throughout the entire study period via the Oura ring.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhosis with clinically significant portal hypertension or decompensation defined by Baveno VII criteria [de Franchis R et al 2022]
* Adults over age 18
* CHE (defined by PHES≤ -4) or previously diagnosed HE
* Disturbed sleep, with Pittsburgh Sleep Quality Index (PSQI) ≥5
* Possession of a "smart phone" with Bluetooth capability and ability to download the Oura application (Apple iOS version 14.0 or greater or Android version 8.0 or higher)

Exclusion Criteria:

* Use of melatonin regularly (3x per week) if unable/unwilling to discontinue for the study
* Inability provide informed consent
* Heavy current alcohol use (>7 drinks weekly for women and 14 drinks weekly for men)'

  -- Body mass index >40
* Known prior sleep disorder including obstructive sleep apnea
* Use of other prescription neuromodulating sleep aides
* Self-reported pregnancy during study screening, as sleep physiology is different in this population

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-08-05 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Mean change in rapid eye movement (REM) sleep as a percentage of total sleep measured by polysomnography after melatonin vs thiamine | Approximately 4 weeks and 9 weeks, at polysomnography which marks the end of each treatment (melatonin or thiamine) assignment.
  Prior research by the investigators and other groups have suggested that patients with hepatic encephalopathy have reduced REM sleep, which is a critical sleep phase that contributes to daytime attention, cognition, and mental/emotional wellbeing. Melatonin has been noted in small studies to increase the amount of nightly REM sleep but is understudied in cirrhosis. The primary outcome of this study will be to determine whether relative to thiamine, use of melatonin increases the absolute nightly amount of REM sleep and the percentage of nightly sleep spent in REM. This outcome will be measured by polysomnography, the gold standard for sleep stage determination..

SECONDARY OUTCOMES:
Mean change in total sleep time measured by polysomnography | Approximately 4 weeks and 9 weeks, at polysomnography which marks the end of each treatment (melatonin or thiamine) assignment.
  The mean difference in individuals in total sleep duration after use of melatonin or thiamine
Mean change in deep sleep time measured by polysomnography | Approximately 4 weeks and 9 weeks, at polysomnography which marks the end of each treatment (melatonin or thiamine) assignment
  The mean difference in individuals in total deep sleep duration and as a percentage of total sleep duration after use of melatonin or thiamine
Mean change in percentage sleep efficiency measured by polysomnography | approximately 4 weeks and 9 weeks, at polysomnography which marks the end of each treatment (melatonin or thiamine) assignment
  The mean difference in individuals in sleep efficiency, as measured by % of total time in bed spent asleep after use of melatonin or thiamine
Mean change in wake after sleep onset (WASO) measured by polysomnography | approximately 4 weeks and 9 weeks, at polysomnography which marks the end of each treatment (melatonin or thiamine) assignment
  The mean difference in individuals in WASO, as measured by duration (min) of wake time after initial sleep onset after use of melatonin or thiamine
Mean change in resting and mean heart rate during sleep measured by polysomnography | approximately 4 weeks and 9 weeks, at polysomnography which marks the end of each treatment (melatonin or thiamine) assignment
  The mean difference in individuals in heart rate (bpm), as measured by average during a whole sleep period and lowest recorded rate after initial sleep onset after use of melatonin or thiamine
Mean change in total sleep time measured by Oura 3.0 | Entire duration of study period (visit 1-3). Approximately week 0-9
  The mean difference in individuals in total sleep duration after use of melatonin or thiamine
Mean change in rapid eye movement (REM) sleep as a percentage of total sleep measured by Oura 3.0 ring after melatonin vs thiamine | Entire duration of study period (visit 1-3). Approximately week 0-9
  Throughout the study, participants will also wear a wearable sleep tracker that is commercially available, the Oura 3.0 ring. This ring performs sleep staging nightly with prior studies suggesting significant agreement with polysomnography, but is inadequately validated against PSG in cirrhosis. REM as a median nightly duration and median percentage of nightly sleep will be measured and compared between each treatment arm for the full 30 day duration.
Mean change in deep sleep time measured by Oura 3.0 | Entire duration of study period (visit 1-3). Approximately week 0-9
  The mean difference in individuals in total deep sleep duration and as a percentage of total sleep duration after use of melatonin or thiamine
Mean change in percentage sleep efficiency measured by Oura 3.0 | Entire duration of study period (visit 1-3). Approximately week 0-9
  The mean difference in individuals in sleep efficiency, as measured by % of total time in bed spent asleep after use of melatonin or thiamine
Mean change in average and resting heart rate during sleep measured by Oura 3.0 | Entire duration of study period (visit 1-3). Approximately week 0-9
  The mean difference in individuals in heart rate (bpm), as measured by average during a whole sleep period after initial sleep onset after use of melatonin or thiamine
Mean change in sleep midpoint as measured by Oura 3.0 | Entire duration of study period (visit 1-3). Approximately week 0-9
  The mean difference in individuals in sleep midpoint (midpoint between sleep onset and awakening) after use of melatonin or thiamine
Variation in sleep midpoint as measured by Oura 3.0 | Entire duration of study period (visit 1-3). Approximately week 0-9
  The mean variability (standard deviation) in individuals in overnight sleep midpoint after use of melatonin or thiamine
Variation in body temperature as measured by Oura 3.0 | Entire duration of study period (visit 1-3). Approximately week 0-9
  The mean variability (standard deviation) in individuals in overnight peripheral body temperature (degrees Celsius) after use of melatonin or thiamine
Mean change in sleep onset time as measured by Oura 3.0 | Entire duration of study period (visit 1-3). Approximately week 0-9
  The mean difference in individuals in sleep onset after use of melatonin or thiamine
Mean change in cognitive performance as measured by Psychometric Hepatic Encephalopathy Score (PHES) | At time of polysomnography (Approximately week 4 and week 9)
  Change in PHES as assessed prior to polysomnography after treatment with melatonin or thiamine. The Psychometric Hepatic Encephalopathy Score (PHES) is a validated, paper-and-pencil neuropsychological battery used to detect minimal or covert hepatic encephalopathy. It evaluates multiple cognitive domains including psychomotor speed, attention, visual perception, and visuomotor coordination.
  Each test is scored and converted to standardized z-scores based on age- and education-adjusted normative data. The total PHES score is the sum of the standardized scores from all five subtests.
  Total scores range from -18 to +6.
  A score of +6 indicates optimal cognitive performance.
  A score of -4 or below is commonly used as the threshold for covert (minimal) hepatic encephalopathy.
Mean difference in subjective sleep quality as measured by Pittsburgh Sleep Quality Index (PSQI) | At time of polysomnography (Approximately week 4 and week 9)
  Change in PSQI as assessed prior to polysomnography after treatment with melatonin or thiamine. The Pittsburgh Sleep Quality Index (PSQI) is a widely used, validated self-report questionnaire that assesses subjective sleep quality over the past month. There are 7 components:
  Subjective sleep quality. Sleep latency, Sleep duration, Habitual sleep efficiency, Sleep disturbances, Use of sleeping medication, Daytime dysfunction
  Each component is scored from 0 (no difficulty) to 3 (severe difficulty), and the component scores are summed to yield a global PSQI score.
  Total scores range from 0 to 21.
  A score of 0 indicates no sleep difficulty, while 21 is severe sleep difficulty
  A score of 5 or greater will be used as a threshold to indicate poor sleep quality.
Mean difference in health related quality of life as measured by PROMIS-29 v2.0 PROPr | At time of polysomnography (Approximately week 4 and week 9)
  Change in PROMIS-29 v2.0 PROPr as assessed prior to polysomnography after treatment with melatonin or thiamine. The PROMIS-29 v2.0 (Patient-Reported Outcomes Measurement Information System 29-item profile, version 2.0) is a standardized health-related quality of life (HRQoL) instrument developed by the NIH. It assesses 7 domains: physical function, anxiety, depression, fatigue, sleep disturbance, ability to participate in social roles and activities, and pain interference, plus a single pain intensity item.
  The PROPr (Preference-Based Scoring System for PROMIS) is a utility score derived from PROMIS domain scores using societal preference weights. It produces a single summary measure of overall health utility suitable for economic evaluations such as quality-adjusted life years (QALYs).
  Total scores range from -0.022 to 1.0.
  A score of 1.0 represents full health.
  A score of 0 represents a health state equivalent to death.
  Scores below 0 (minimum -0.022) indicate health states con
Mean change in pre-bedtime to awake salivary melatonin levels in participants after 4 weeks of treatment with melatonin or thiamine as measured at time of polysomnography | At time of polysomnography (Approximately week 4 and week 9)
  We will collect night and morning salivary melatonin levels and assess the difference between the two levels after each treatment period. The mean change in melatonin levels will be compared between the two treatment assignments.
Correlation in measurement of deep sleep determination between polysomnography and Oura 3.0 ring | Entire time of concomitant measurement with both devices (Oura/PSG), which is during each polysomnography, approximately weeks 4 and 9.
  Both Oura and polysomnography assess sleep phases (awake, light sleep, deep sleep and REM sleep) on an epoch (5 minutes for Oura, one minute for polysomnography) level. We will assess intraclass coefficient and generate Bland-Altman plots for agreement between Oura and polysomnography on deep sleep stage
Correlation in measurement of light sleep determination between polysomnography and Oura 3.0 ring | Entire time of concomitant measurement with both devices (Oura/PSG), which is during each polysomnography, approximately weeks 4 and 9.
  Both Oura and polysomnography assess sleep phases (awake, light sleep, deep sleep and REM sleep) on an epoch (5 minutes for Oura, one minute for polysomnography) level. We will assess intraclass coefficient and generate Bland-Altman plots for agreement between Oura and polysomnography on light sleep stage
Correlation in measurement of rapid eye movement (REM) sleep determination between polysomnography and Oura 3.0 ring | Entire time of concomitant measurement with both devices (Oura/PSG), which is during each polysomnography, approximately weeks 4 and 9.
  Both Oura and polysomnography assess sleep phases (awake, light sleep, deep sleep and REM sleep) on an epoch (5 minutes for Oura, one minute for polysomnography) level. We will assess intraclass coefficient and generate Bland-Altman plots for agreement between Oura and polysomnography on REM sleep stage
Correlation in measurement of awake/sleep determination between polysomnography and Oura 3.0 ring | Entire time of concomitant measurement with both devices (Oura/PSG), which is during each polysomnography, approximately weeks 4 and 9.
  Both Oura and polysomnography assess sleep phases (awake, light sleep, deep sleep and REM sleep) on an epoch (5 minutes for Oura, one minute for polysomnography) level. We will assess intraclass coefficient and generate Bland-Altman plots for agreement between Oura and polysomnography on sleep vs awake.
Correlation in measurement of heart rate between polysomnography and Oura 3.0 ring | Entire time of concomitant measurement with both devices (Oura/PSG), which is during each polysomnography, approximately weeks 4 and 9.
  Both Oura and polysomnography assess mean heart rate on an epoch (60 second) level. We will assess intraclass coefficient and generate Bland-Altman plots for agreement between Oura and polysomnography on heart rate measurement

CONTACTS AND LOCATIONS:
Overall Officials: Adam Buckholz, MD MS, Principal Investigator — NewYork-Presbyterian/Weill Cornell Medical College
Locations (1):
- NewYork-Presbyterian/Weill Cornell Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
de-identified study data that underlie results in a publication.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication
Access Criteria: Researchers who provide a methodologically sound proposal, to achieve aims in the approved proposal. Proposals should be directed to apb9012@med.cornell.edu. To gain access, data requestors will need to sign a data access agreement. Data will be available for 5 years after publication at a third party website.

REFERENCES:
- [Background] de Zambotti M, Rosas L, Colrain IM, Baker FC. The Sleep of the Ring: Comparison of the OURA Sleep Tracker Against Polysomnography. Behav Sleep Med. 2019 Mar-Apr;17(2):124-136. doi: 10.1080/15402002.2017.1300587. Epub 2017 Mar 21. PMID 28323455
- [Background] Desai AP, Madathanapalli A, Tang Q, Orman ES, Lammert C, Patidar KR, Nephew LD, Ghabril M, Monahan PO, Chalasani N. PROMIS Profile-29 is a valid instrument with distinct advantages over legacy instruments for measuring the quality of life in chronic liver disease. Hepatology. 2023 Dec 1;78(6):1788-1799. doi: 10.1097/HEP.0000000000000480. Epub 2023 May 25. PMID 37222262
- [Background] Tapper EB, Lai JC. Time to embrace PROMIS-29 as the standard health-related quality of life instrument for patients with cirrhosis. Hepatology. 2023 Dec 1;78(6):1688-1691. doi: 10.1097/HEP.0000000000000508. Epub 2023 Jun 7. No abstract available. PMID 37278246
- [Background] Wellek S, Blettner M. On the proper use of the crossover design in clinical trials: part 18 of a series on evaluation of scientific publications. Dtsch Arztebl Int. 2012 Apr;109(15):276-81. doi: 10.3238/arztebl.2012.0276. Epub 2012 Apr 13. PMID 22567063
- [Background] Enezi AAl, Al-Jahdali F, Ahmed AE, Shirbini N, Harbi AAl, Salim B, Ali YZ, Abdulrahman A, Khan M, Khaleid A, Hamdan AJ. Symptoms of Daytime Sleepiness and Sleep Apnea in Liver Cirrhosis Patients. Ann Hepatol. 2017 Jul-Aug;16(4):591-598. doi: 10.5604/01.3001.0010.0304. PMID 28611264
- [Background] de Franchis R, Bosch J, Garcia-Tsao G, Reiberger T, Ripoll C; Baveno VII Faculty. Baveno VII - Renewing consensus in portal hypertension. J Hepatol. 2022 Apr;76(4):959-974. doi: 10.1016/j.jhep.2021.12.022. Epub 2021 Dec 30. PMID 35120736
- [Background] Weissenborn K. Hepatic Encephalopathy: Definition, Clinical Grading and Diagnostic Principles. Drugs. 2019 Feb;79(Suppl 1):5-9. doi: 10.1007/s40265-018-1018-z. PMID 30706420
- [Background] Ghabril M, Jackson M, Gotur R, Weber R, Orman E, Vuppalanchi R, Chalasani N. Most Individuals With Advanced Cirrhosis Have Sleep Disturbances, Which Are Associated With Poor Quality of Life. Clin Gastroenterol Hepatol. 2017 Aug;15(8):1271-1278.e6. doi: 10.1016/j.cgh.2017.01.027. Epub 2017 Feb 3. PMID 28167158
- [Background] De Silva AP, Niriella MA, Ediriweera DS, De Alwis JP, Liyanage IK, Ettickan U, Liyanapathirana KV, Undugodage C, de Silva HA, de Silva HJ. Low-dose melatonin for sleep disturbances in early-stage cirrhosis: A randomized, placebo-controlled, cross-over trial. JGH Open. 2020 May 18;4(4):749-756. doi: 10.1002/jgh3.12356. eCollection 2020 Aug. PMID 32782966
- [Background] Almeida Montes LG, Ontiveros Uribe MP, Cortes Sotres J, Heinze Martin G. Treatment of primary insomnia with melatonin: a double-blind, placebo-controlled, crossover study. J Psychiatry Neurosci. 2003 May;28(3):191-6. PMID 12790159
- [Background] Cajochen C, Krauchi K, Mori D, Graw P, Wirz-Justice A. Melatonin and S-20098 increase REM sleep and wake-up propensity without modifying NREM sleep homeostasis. Am J Physiol. 1997 Apr;272(4 Pt 2):R1189-96. doi: 10.1152/ajpregu.1997.272.4.R1189. PMID 9140019
- [Background] Kunz D, Mahlberg R, Muller C, Tilmann A, Bes F. Melatonin in patients with reduced REM sleep duration: two randomized controlled trials. J Clin Endocrinol Metab. 2004 Jan;89(1):128-34. doi: 10.1210/jc.2002-021057. PMID 14715839
- [Background] Montagnese S, Middleton B, Mani AR, Skene DJ, Morgan MY. Sleep and circadian abnormalities in patients with cirrhosis: features of delayed sleep phase syndrome? Metab Brain Dis. 2009 Sep;24(3):427-39. doi: 10.1007/s11011-009-9146-5. PMID 19756996
- [Background] Boeve BF, Silber MH, Ferman TJ. Melatonin for treatment of REM sleep behavior disorder in neurologic disorders: results in 14 patients. Sleep Med. 2003 Jul;4(4):281-4. doi: 10.1016/s1389-9457(03)00072-8. PMID 14592300
- [Background] Chinoy ED, Cuellar JA, Huwa KE, Jameson JT, Watson CH, Bessman SC, Hirsch DA, Cooper AD, Drummond SPA, Markwald RR. Performance of seven consumer sleep-tracking devices compared with polysomnography. Sleep. 2021 May 14;44(5):zsaa291. doi: 10.1093/sleep/zsaa291. PMID 33378539
- [Background] Depner CM, Cheng PC, Devine JK, Khosla S, de Zambotti M, Robillard R, Vakulin A, Drummond SPA. Wearable technologies for developing sleep and circadian biomarkers: a summary of workshop discussions. Sleep. 2020 Feb 13;43(2):zsz254. doi: 10.1093/sleep/zsz254. PMID 31641776
- [Background] Malhotra A, Younes M, Kuna ST, Benca R, Kushida CA, Walsh J, Hanlon A, Staley B, Pack AI, Pien GW. Performance of an automated polysomnography scoring system versus computer-assisted manual scoring. Sleep. 2013 Apr 1;36(4):573-82. doi: 10.5665/sleep.2548. PMID 23565003
- [Background] Marjot T, Ray DW, Williams FR, Tomlinson JW, Armstrong MJ. Sleep and liver disease: a bidirectional relationship. Lancet Gastroenterol Hepatol. 2021 Oct;6(10):850-863. doi: 10.1016/S2468-1253(21)00169-2. Epub 2021 Jul 15. PMID 34273289
- [Background] Bajaj JS, Saeian K, Schubert CM, Franco R, Franco J, Heuman DM. Disruption of sleep architecture in minimal hepatic encephalopathy and ghrelin secretion. Aliment Pharmacol Ther. 2011 Jul;34(1):103-5. doi: 10.1111/j.1365-2036.2011.04681.x. No abstract available. PMID 21631553
- [Background] Buckholz A, Clarke L, Paik P, Jesudian A, Schwartz R, Krieger A, Rosenblatt R, Brown RS Jr. Evaluating sleep in covert encephalopathy with wearable technology: results from the WATCHES study. Hepatol Commun. 2023 Feb 1;7(2):e0002. doi: 10.1097/HC9.0000000000000028. eCollection 2023 Feb 1. PMID 36724117
- [Background] Liu C, Zhou J, Yang X, Lv J, Shi Y, Zeng X. Changes in sleep architecture and quality in minimal hepatic encephalopathy patients and relationship to psychological dysfunction. Int J Clin Exp Med. 2015 Nov 15;8(11):21541-8. eCollection 2015. PMID 26885103
- [Background] Labenz C, Baron JS, Toenges G, Schattenberg JM, Nagel M, Sprinzl MF, Nguyen-Tat M, Zimmermann T, Huber Y, Marquardt JU, Galle PR, Worns MA. Prospective evaluation of the impact of covert hepatic encephalopathy on quality of life and sleep in cirrhotic patients. Aliment Pharmacol Ther. 2018 Aug;48(3):313-321. doi: 10.1111/apt.14824. Epub 2018 Jun 4. PMID 29863286
- [Background] Steindl PE, Finn B, Bendok B, Rothke S, Zee PC, Blei AT. Disruption of the diurnal rhythm of plasma melatonin in cirrhosis. Ann Intern Med. 1995 Aug 15;123(4):274-7. doi: 10.7326/0003-4819-123-4-199508150-00005. PMID 7611593
- [Background] Bersagliere A, Raduazzo ID, Nardi M, Schiff S, Gatta A, Amodio P, Achermann P, Montagnese S. Induced hyperammonemia may compromise the ability to generate restful sleep in patients with cirrhosis. Hepatology. 2012 Mar;55(3):869-78. doi: 10.1002/hep.24741. Epub 2012 Jan 19. PMID 21994139
- [Background] SHERLOCK S, SUMMERSKILL WH, WHITE LP, PHEAR EA. Portal-systemic encephalopathy; neurological complications of liver disease. Lancet. 1954 Sep 4;267(6836):454-7. No abstract available. PMID 13193045
- [Background] Tapper EB, Halbert B, Mellinger J. Rates of and Reasons for Hospital Readmissions in Patients With Cirrhosis: A Multistate Population-based Cohort Study. Clin Gastroenterol Hepatol. 2016 Aug;14(8):1181-1188.e2. doi: 10.1016/j.cgh.2016.04.009. Epub 2016 Apr 13. PMID 27085758
- [Background] Lauridsen MM, Bajaj JS. Hepatic encephalopathy treatment and its effect on driving abilities: A continental divide. J Hepatol. 2015 Jul;63(1):287-8. doi: 10.1016/j.jhep.2015.03.017. Epub 2015 Mar 18. No abstract available. PMID 25796480
- [Background] Bajaj JS, Heuman DM, Sterling RK, Sanyal AJ, Siddiqui M, Matherly S, Luketic V, Stravitz RT, Fuchs M, Thacker LR, Gilles H, White MB, Unser A, Hovermale J, Gavis E, Noble NA, Wade JB. Validation of EncephalApp, Smartphone-Based Stroop Test, for the Diagnosis of Covert Hepatic Encephalopathy. Clin Gastroenterol Hepatol. 2015 Oct;13(10):1828-1835.e1. doi: 10.1016/j.cgh.2014.05.011. Epub 2014 May 17. PMID 24846278
- [Background] European Association for the Study of the Liver. EASL Clinical Practice Guidelines on the management of hepatic encephalopathy. J Hepatol. 2022 Sep;77(3):807-824. doi: 10.1016/j.jhep.2022.06.001. Epub 2022 Jun 17. PMID 35724930
- [Background] Hartmann IJ, Groeneweg M, Quero JC, Beijeman SJ, de Man RA, Hop WC, Schalm SW. The prognostic significance of subclinical hepatic encephalopathy. Am J Gastroenterol. 2000 Aug;95(8):2029-34. doi: 10.1111/j.1572-0241.2000.02265.x. PMID 10950053
- [Background] Ridola L, Cardinale V, Riggio O. The burden of minimal hepatic encephalopathy: from diagnosis to therapeutic strategies. Ann Gastroenterol. 2018 Mar-Apr;31(2):151-164. doi: 10.20524/aog.2018.0232. Epub 2018 Feb 1. PMID 29507462